CLINICAL TRIAL: NCT07339111
Title: Randomized, Prospective, Double Blind, Multi-Center, Phase 3 Pivotal Clinical Trial to Compare Efficacy and Safety of CARTISTEM® and Surgical Comparator in Subjects With Knee Cartilage Lesions and Osteoarthritis
Brief Title: Phase 3 Pivotal Trial Comparing CARTISTEM® and Surgical Comparator for Knee Cartilage Lesions and Osteoarthritis
Acronym: CARTISTEM23-01
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medipost, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPA-CARTISTEM-2023-01
Record Dates: First submitted 2026-01-09; First posted 2026-01-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Knee Cartilage Defects
Keywords: symptomatic knee cartilage defects; knee cartilage; cartilage repair; osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Debridement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CARTISTEM + Debridement (Experimental): Participants in Group A will receive CARTISTEM + Debridement in the target knee.
  Interventions: Biological: CARTISTEM® + Debridement
- Debridement (Active Comparator): Participants in Group B will receive debridement procedure.
  Interventions: Procedure: Debridement

INTERVENTIONS:
Biological: CARTISTEM® + Debridement — CARTISTEM® + Debridement
  CARTISTEM® consists of approximately 7.5 x 106 hUCB-MSCs (human umbilical cord blood-derived mesenchymal stem/stromal cells) suspended in 1.5 ml medium in one vial, and 60 mg sodium hyaluronate provided as a lyophilized powder in a separate vial.
  A viscous and malleable gel matrix is formed by mixing hUCB-MSCs (main component) and 60mg of sodium hyaluronate at a 4% concentration (excipient).
  Arms: CARTISTEM + Debridement
Procedure: Debridement — Debridement of unstable cartilage in and around cartilage lesion(s) in the knee.
  Arms: Debridement

SUMMARY:
To establish the efficacy and safety of CARTISTEM®, a combination product composed of allogeneic human umbilical cord blood-derived mesenchymal stem cells (hUCB-MSCs) formulated with a cross-linked sodium hyaluronate (HA) hydrogel, CARTISTEM® compared to the surgical comparator of debridement in Subjects with knee cartilage lesions and osteoarthritis.

This trial is intended to provide evidence of the superiority of CARTISTEM® to reduce knee pain and improve knee function compared to debridement for Subjects with knee cartilage lesions and osteoarthritis at 2-years post-treatment.

Additionally, this trial is intended to intended to explore whether CARTISTEM® may have disease-modifying effects on osteoarthritis progression through the use of semi-quantitative MRI assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years old.
2. Knee Osteoarthritis diagnosed in the index knee according to the clinical definition of American College of Rheumatology (ACR) guidelines at screening.
3. Failed conservative knee osteoarthritis treatment for at least 3 months prior to consent (weight reduction, physical therapy, injections, pain medications, etc.).
4. Kellgren-Lawrence (KL) in the index knee of grade 2 to 3 as determined by independent radiologist review of study X-Ray.
5. Clinically relevant femoral cartilage defects classified using modified Outerbridge Grade 3 or 4 in index knee with combined lesion area ≥ 2 cm2 and ≤ 9 cm2 and at least a single femoral lesion ≥ 2 cm2 as determined by independent radiologist review of study MRI.
6. Body Mass Index (BMI) ≤ 35 kg / m2 .
7. VAS PAIN index knee score ≥ 40 to ≤ 90 based on 100-point scale at screening.
8. VAS PAIN contralateral knee score ≤ 30 based on 100-point scale at screening.
9. WOMAC® FUNCTION index knee mean score ≥ 25 to ≤ 90 based on 100-point scale at screening.
10. WOMAC® Pain index knee mean score ≥ 40 to ≤ 90 based on 100-point VAS (visual analogue scale) at screening.
11. Subjects must be willing to abstain from treatments in the index knee from the time the informed consent is signed until after the last study follow up visit.
12. Subjects must be willing to discontinue analgesics except:

    * Rescue medication (acetaminophen) allowed for break-through pain throughout the study.
    * Subjects must be willing to discontinue use of all pain medications at least 48 hours prior to baseline assessment and each follow up visit.
    * Limited postoperative NSAID use is permissible per IND clinical guidance and site manual, provided washout before scheduled efficacy assessments.
    * Post operative narcotics.
13. Subjects with stage 3 hypertension (systolic ≥ 180 mm Hg and diastolic ≥ 120 mmHg) must have blood pressure (BP) controlled prior to surgical procedure.
14. Subject's central lab results are within normal ranges or deemed as not clinically significant by investigator for CARTISTEM® treatment or surgical comparator.
15. Female Subjects of childbearing potential must agree to practice adequate methods of birth control to prevent pregnancy during the study.
16. Subjects must be able to comply fully with the rehabilitation requirements.
17. Subjects must be able to understand and comply with the requirements of the study.
18. Subjects must voluntarily provide written informed consent.

Exclusion Criteria:

1. Subject received an IA injection of Hyaluronic Acid (HA), Platelet Rich Plasma (PRP), Bone Marrow Aspirate / Concentrate (BMA / BMAC), long-acting / conventional steroid, or investigational drug in either knee within 3 months of signing informed consent. Note: injections of the contralateral knee are allowed during the trial.
2. Bone marrow lesion (BML) grade 3 on femur, tibia, or patella except at femoral lesion area (BML grade 3 allowed) in index knee as determined by independent radiologist review of study MRI.
3. KL index knee grade 0, 1 or 4 as determined by independent radiologist review of study X-Ray.
4. KL Contralateral knee severity grade 4 as determined by independent radiologist review of study X-Ray.
5. Anatomical axis varus or valgus malalignment ≥ 6° in either knee as determined by independent radiologist.
6. Joint ligament instability in index knee ≥ Grade 3 or ligament instability that would require surgical intervention as determined by investigator or designee.
7. Complete meniscal deficiency, meniscal root tears and / or severe meniscal extrusion as determined by independent radiologist.
8. Kissing bipolar lesions (tibial or patellar) Outerbridge 4 exceeding 25% of the femoral lesion area in size and/or penetrating through the subchondral bone as determined by independent radiologist.
9. Surgery of the index knee joint within 6 months of signing the informed consent. Investigator confirms that Subject has recovered from any prior surgical intervention to enable treatment within this study protocol. No radiation therapy of the index knee as determined by documented medical history.
10. Chronic inflammatory articular diseases such as rheumatoid arthritis, gout, pseudogout, gouty arthritis, or fibromyalgia as determined by documented medical history.
11. Bone disorders of index knee: osteonecrosis including avascular necrosis (AVN); Osteochondritis dissecans (OCD); Spontaneous Osteonecrosis of the Knee (SONK); Subchondral Insufficiency Fracture (SIF); Subchondral / intraosseous bone cyst >4mm at femoral treatment location, bone tumors, bone contusion or stress fracture, pathologic fracture, and other bone exclusionary findings as determined by independent radiologist review of study MRI or X-ray.
12. Joint disorders of the index knee including infection, osteomyelitis, soft tissue tumors, and bone marrow infiltration as determined by independent radiologist review of study MRI or X-ray.
13. Diseases or disorders including Paget's disease, ochronosis, acromegaly, haemochromatosis, Wilson's disease, genetic disease (hyperkinesia, etc.), or genetic collagen disorder as determined by documented medical history.
14. Vascular or neurological disorders of the lower extremities as determined by documented medical history. Note: Varicose veins are not an exclusion criteria.
15. Autoimmune diseases - documented medical history. Addison's Disease, Dermatomyositis, Irritable Bowel Diseases (IBD) or Irritable Bowel Syndrome (IBS) (including Crohn's disease and ulcerative colitis), Multiple sclerosis, Myasthenia gravis, Pernicious anemia, Rheumatoid Arthritis, Sjogren's Syndrome, systemic Lupus erythematosus. Note: Celiac disease is not an exclusion criterion.
16. Subject has documented systemic diseases such as but not limited to HIV, hepatitis, HTVL, syphilis, and blood coagulopathies (including hemophilia, Von Willebrand disease, thrombocytopenia, disseminated intravascular coagulation (DIC)). Note: Occurrence of Deep Vein Thrombosis ≥ 5 years prior to consent is not an exclusion.
17. Subject is taking anticoagulant medication (e.g., warfarin, (Coumadin), apixaban (Eliquis), rivaroxaban (Xarelto), clopidogrel (Plavix) or equivalent) but not excluding 81mg aspirin.
18. Uncontrolled diabetes with HbA1c > 8% as determined by documented medical history.
19. Infectious disease requiring parenteral administration of antibiotics.
20. Administered immunosuppressants such as Cyclosporin A or azathioprine within 6 months of signing the informed consent.
21. Subject has received chemotherapy in the 12 months prior to signing informed consent.
22. Subject has received other allogeneic stem cell therapy.
23. Prior cartilage repair procedure (such as MACI, ACI, OATS, OCA, Agili-C) in the index knee or the index knee contains a uni-compartmental knee replacement. Revision of a prior microfracture procedure is allowed if subchondral plate remains intact and lesion is lacking significant intra-lesional osteophytes.
24. Prior invasive knee osteoarthritis treatment including subchondroplasty, cryoneurolysis, genicular nerve ablation, genicular artery embolization, in situ MISHA (medial knee implanted shock absorber), prosthetic implants or other knee implants or invasive treatments for the index knee.
25. Known history of hypersensitivity / allergy to hyaluronan.
26. Currently pregnant or nursing.
27. Psychotic diseases, epilepsy, or any history of such diseases.
28. Known substance or alcohol abuse in the prior 3 years.
29. Contraindication to MRI imaging or unwillingness to undergo MRI.
30. Currently receiving or in litigation related to workman's compensation, personal injury, or disability claims.
31. Considered by principal investigator inappropriate for the clinical trial due to any reasons other than those listed above.

Baseline PRO Assessment Inclusion Criteria:

1. VAS PAIN index knee score ≥ 40 to ≤ 90 based on 100-point scale at baseline PRO assessment.
2. WOMAC® FUNCTION index knee mean score ≥ 25 to ≤ 90 based on 100-point scale at baseline PRO assessment.

Baseline Surgical Inclusion Criteria:

1. Treated cartilage defects Outerbridge Grade 3 or 4 in index knee with combined femoral lesion area ≤ 9 cm2 as determined arthroscopically or by arthrotomy by treating physician.

Baseline Surgical Exclusion Criteria:

1. Meniscal root tears and / or severe meniscal extrusion or non-functional meniscus as determined arthroscopically or by arthrotomy by treating physician.
2. Kissing bipolar lesions (tibial or patellar) Outerbridge 4 exceeding 25% of the femoral lesion area in size and/or penetrating through the subchondral bone as determined arthroscopically or by arthrotomy by treating physician.
3. Bone or joint disorders of the index knee including infection, osteomyelitis, soft tissue tumors, bone marrow infiltration, osteonecrosis (AVN or OCD) as determined arthroscopically or by arthrotomy by treating physician.
4. Identification of prior cartilage repair procedure (such as MACI, ACI, OATS, OCA, Agili-C) or uni-compartmental knee replacement in the index knee as determined arthroscopically or by arthrotomy by treating physician. Revision of a prior microfracture procedure is allowed if subchondral bone remains intact and lacking significant intra-lesional osteophytes.
5. Subject is documented as pregnant based on hCG urine or blood test prior to surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain Score | From enrollment to end of follow-up at 24 months
  Change from Baseline Visual Analog Scale (VAS) Pain score (0-100 point scale, 0 being no pain at one end and 100 being the worst imaginable pain at the other) in index knee comparing CARTISTEM® to surgical control at 24-months post-treatment.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC®) Function score | From start of treatment to the end of follow-up at 24 months
  Change from Baseline Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC®) Function score (0-100 point scale, 0 being the best functioning and 100 being the worst functioning) in index knee comparing CARTISTEM® to surgical control at 24-months post-treatment.

SECONDARY OUTCOMES:
Modified Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) Score | enrollment to follow-up at 24 months.
  Change in modified MOCART score in Index knee comparing CARTISTEM® to surgical control at 24-months post-treatment.
Change in MRI Osteoarthritis Knee Score (MOAKS) cartilage morphology | enrollment to follow up at 24 months
  Change in MOAKS cartilage morphology with delta sum score - extent of cartilage damage score in Index knee comparing CARTISTEM® to surgical control at 24-months post-treatment.

OTHER OUTCOMES:
Change in Western Ontario and McMaster Universities OA Index (WOMAC®) Total score (0-100 point scale, 0 being no osteoarthritis symptoms and 100 being the worst symptoms) in index knee comparing CARTISTEM® to surgical control at 24-months post-treatment. | enrollment to follow up at 24 months
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC®) Stiffness score (0-100 point scale, 0 being the no stiffness, 100 being the most) in index knee comparing CARTISTEM® to surgical control at 24-months post-treatment. | enrollment to follow up at 24 months
Change in EuroQoL 5 Dimensions, 5 Levels (5D-5L, with 0 being the worst and 100 being the best) comparing CARTISTEM® to surgical control at 24-months post-treatment. | enrollment at follow up at 24 months
Change in MOAKS intercondylar synovitis comparing CARTISTEM® to surgical control at 24-months post-treatment. | enrollment to follow up at 24 months
Change in MOAKS whole knee effusion comparing CARTISTEM® to surgical control at 24-months post-treatment. | enrollment to follow up at 24 months
Change in MRI Osteoarthritis Knee Score (MOAKS) cartilage morphology - extent of cartilage damage comparing CARTISTEM® to surgical control at 24-months post-treatment | Enrollment to follow up at 24 months
Change in Evaluator Global Assessment (0-100, 0 being very well, 100 being very poor) comparing CARTISTEM® to surgical control at 24-months post-treatment. | Enrollment to follow up at 24 months
Change in Patient Global Assessment (0-100, 0 being very well, 100 being very poor) comparing CARTISTEM® to surgical control at 24-months post-treatment. | Enrollment to follow up at 24 months.
OMERACT-OARSI responder rate comparing CARTISTEM® to surgical control at 24-months post-treatment. | Enrollment to follow up at 24 months
Treatment failure rate comparing CARTISTEM® to surgical control at 24-months post-treatment. | Enrollment to follow up at 24 months

IPD SHARING:
Plan to Share IPD: No